CLINICAL TRIAL: NCT06636201
Title: Deputy Director of Department of Neurosurgery, the Second Affiliated Hospital of Zhejiang University School of Medicine；Professor；
Brief Title: Large-scale Multi-omics Analysis of Cerebrospinal Fluid
Status: Recruiting | Type: Observational
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Other Study IDs: 2024-0969
Record Dates: First submitted 2024-08-25; First posted 2024-10-10 (Actual); Last update posted 2024-10-10 (Actual); Status verified 2024-08

CONDITIONS: Aging
Keywords: biomarker; aging; neurodegenerative disease
MeSH Terms: conditions — Neurodegenerative Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — cerebrospinal fluid
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The aim of this study is to explore the role of cerebrospinal fluid (CSF) biomarkers in aging and neurodegenerative diseases.

DETAILED DESCRIPTION:
This study aims to investigate the role of cerebrospinal fluid (CSF) biomarkers in aging and neurodegenerative diseases, with a focus on the following objectives:

Analysis of Age-Related Changes in CSF Biomarkers: The study will analyze CSF samples from different age groups to identify biomarkers that undergo significant changes during the aging process. This includes the investigation of amyloid-beta (Aβ42), Tau proteins (including the phosphorylated form p-tau181), and other proteins related to neuroinflammation and blood-brain barrier function.

Development of a Predictive Model for Early Diagnosis: By categorizing and quantifying CSF proteins across various age groups, the study aims to establish a predictive model for the early diagnosis of neurodegenerative diseases, such as Alzheimer's disease. The ability to detect these diseases before clinical symptoms emerge could enable early intervention and treatment, offering a crucial window for therapeutic strategies.

Investigation of Dynamic Changes in CSF Biomarkers Across Disease Stages: The study will examine the dynamic changes in CSF biomarkers at different stages of neurodegenerative diseases, including early, middle, and late stages. Understanding the role of these biomarkers in disease progression will provide insights into the pathological processes and potential therapeutic windows.

Creation of a Comprehensive CSF Biomarker Database: A database will be established, encompassing CSF biomarkers from various age groups, disease states, and treatment responses. This resource will be invaluable for future research, facilitating the scientific community's understanding of neurodegenerative diseases and the development of new therapeutic approaches.

Through the achievement of these objectives, this study aims to advance the application of CSF biomarkers in neuroscience research and clinical practice, ultimately improving the diagnosis, management, and treatment of aging-related and neurodegenerative conditions.

ELIGIBILITY:
1. Inclusion Criteria:

   * Patients aged 0 to 90 years will be selected for the study.
   * Patients admitted for surgery under spinal anesthesia due to non-neurological conditions, such as lower limb fractures or hemorrhoids.
   * Pediatric patients undergoing surgical treatment for tethered spinal cord syndrome.
2. Exclusion Criteria:

   * Patients with neurological conditions, including encephalitis, Parkinson's disease, Alzheimer's disease, hydrocephalus, brain tumors, and psychiatric disorders.

Ages: 0 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Patients admitted for spinal anesthesia surgery due to non-neurological conditions and pediatric patients undergoing surgery for tethered spinal cord syndrome.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2024-03-01 (Actual); Primary Completion 2025-03-01 (Estimated); Study Completion 2025-04-01 (Estimated)

PRIMARY OUTCOMES:
Cerebrospinal fluid (CSF) biomarkers | December 2024
  CSF samples from different ages were analyzed to identify biomarkers that change significantly during aging, such as amyloid beta (Aβ42), Tau protein (including the phosphorylated form p-tau181), and other proteins associated with neuroinflammation and blood-brain barrier function

CONTACTS AND LOCATIONS:
Locations (1):
- The Second Affiliated Hospital, Zhejiang University School of Medicine, Hangzhou, Zhejiang, China

DOCUMENTS (2):
  • Study Protocol (2024-06-27): https://cdn.clinicaltrials.gov/large-docs/01/NCT06636201/Prot_000.pdf
  • Informed Consent Form (2024-06-27): https://cdn.clinicaltrials.gov/large-docs/01/NCT06636201/ICF_001.pdf